CLINICAL TRIAL: NCT02276482
Title: Phase 3 Study of IV to Oral 6-Day Tedizolid Phosphate Compared With 10-day Comparator in Subjects 12 to < 18 Years With cSSTI.
Brief Title: Study of Tedizolid Phosphate in Adolescents With Complicated Skin and Soft Tissue Infection (cSSTI) (MK-1986-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1986-012; TR701-122 (Other: Cubist Pharmaceuticals LLC Protocol Number); 2014-004023-40 (EudraCT Number); MK-1986-012 (Other: Merck)
Record Dates: First submitted 2014-10-09; First posted 2014-10-28 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Skin Diseases, Infectious; Skin Diseases, Bacterial
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial | interventions — tedizolid phosphate; Vancomycin; Cefazolin; Cephalexin; Aztreonam; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tedizolid Phosphate (Experimental): Tedizolid Phosphate IV and/or oral 200 mg once per day for 6 days. Participants with gram-negative wound infection may receive aztreonam (IV) and/or metronidazole (IV or oral).
  Interventions: Drug: Tedizolid Phophate; Drug: Aztreonam; Drug: Metronidazole
- Antibiotic comparator drug (Active Comparator): IV and/or oral antibiotic comparator drug for 10 days. Participants with gram-negative wound infection may receive aztreonam (IV) and/or metronidazole (IV or oral).
  Interventions: Drug: Antibiotic comparator; Drug: Aztreonam; Drug: Metronidazole

INTERVENTIONS:
Drug: Tedizolid Phophate — Tedizolid Phophate 200 mg, IV and/or oral for 6 days
  Other Names: TR701-122; MK-1986; SIVEXTRO®
  Arms: Tedizolid Phosphate
Drug: Antibiotic comparator — Antibiotic comparator drug, IV and/or orally for 10 days. Antibiotic comparator included the following: Vancomycin, Linezolid, Clindamycin, Flucloxacillin, Cefazolin, Cephalexin.
  Other Names: Vancomycin: Vancocin, Firvanq, Lyphocin; Linezolid: Zyvox; Clindamycin: Cleocin; Flucloxacillin: Floxapen, Flopen, Staphylex; Cefazolin: Ancef, Kefzol; Cephalexin: Keflex, Zartan, Panixine, Biocef
  Arms: Antibiotic comparator drug
Drug: Aztreonam — In countries and/or sites where aztreonam is available, adjunctive aztreonam (IV) may be initiated on Day 1 or during the first 3 days of treatment if the participant is determined or suspected to have an infection with gram-negative aerobic pathogens.
  Other Names: Azactam, Cayston
Drug: Metronidazole — Metronidazole (IV or oral) may be initiated on Day 1 or during the first 3 days of treatment if the participant is determined or suspected to have an infection with anaerobic pathogens.
  Other Names: Flagyl, Metro

SUMMARY:
The purpose of the study is to compare the safety of intravenous (IV) and/or oral 6-day 200 mg tedizolid phosphate with 10-day comparator in participants 12 to <18 years with cSSTI.

DETAILED DESCRIPTION:
A randomized, single-blind, multicenter, Phase 3 study of IV and/or oral tedizolid phosphate 200 mg once per day for 6 days compared with IV and/or oral comparator for 10 days for the treatment of cSSTI, also known as acute bacterial skin and skin structure infections, in participants 12 to <18 years. cSSTI includes major cutaneous abscess, cellulitis/erysipelas, and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 years to <18 years
* Adequate venous access for IV administration of study drug for at least 24 hours (for participants receiving IV medication) and collection of protocol-specified blood samples
* Local symptoms must have started within 7 days before Study Day -1
* cSSTI meeting at least 1 of the clinical syndrome definitions.
* Suspected or documented Gram-positive infection from baseline Gram stain or culture.
* Parent/legally authorized representative (LAR) able to give informed consent and willing and able to comply with all required study procedures. Assent is also required of children who in the Investigator's judgment are capable of understanding the nature of the study

Exclusion Criteria:

* Uncomplicated minor skin and skin structure infections such as pustules, folliculitis, furuncles, minor abscesses (small volume of suppuration not surrounded by cellulitis/erysipelas), impetiginous lesions, superficial or limited cellulitis/erysipelas, and minor wound associated foreign body reactions (eg, stitch abscesses)
* Known bacteremia, severe sepsis or septic shock
* Recent history of opportunistic infections where the underlying cause of these infections is still active (eg, leukemia, transplant, acquired immunodeficiency syndrome)
* Hypersensitivity to tedizolid phosphate or any component in the formulation
* Hypersensitivity to all of the comparator drugs; hypersensitivity to a comparator drug does not preclude participation if an alternative comparator can be used
* For participants with wound infections: history of hypersensitivity to ceftazidime, aztreonam, or any component of the aztreonam formulation, if aztreonam adjunctive therapy is required; history of hypersensitivity to metronidazole or any component of the formulation, if metronidazole adjunctive therapy is required
* Needs oral administration of methotrexate, topotecan, irinotecan or rosuvastatin, during administration of oral study drug.
* Uses monoamine oxidase inhibitors, tricyclic antidepressants, buspirone, selective serotonin reuptake inhibitors and serotonin 5 hydroxytryptamine receptor agonists (triptans) within 14 days prior to study drug administration

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bradley JS, Antadze T, Ninov B, Tayob MS, Broyde N, Butterton JR, Chou MZ, De Anda CS, Kim JY, Sears PS. Safety and Efficacy of Oral and/or Intravenous Tedizolid Phosphate From a Randomized Phase 3 Trial in Adolescents With Acute Bacterial Skin and Skin Structure Infections. Pediatr Infect Dis J. 2021 Mar 1;40(3):238-244. doi: 10.1097/INF.0000000000003010. PMID 33395210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who were enrolled and provided informed consent/ascent were randomized to one of two treatment groups.
Period: Overall Study
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Started | 91 | 29
Completed | 88 | 28
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Gram-negative infection | 1 | 0
Not completed — Reason not specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug | Total
Number analyzed (Participants) | 91 | 29 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.4 (1.7) | 14.4 (2.0) | 14.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 12 | 45
  Male | 58 | 17 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 86 | 28 | 114
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 80 | 24 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events on Tedizolid Phosphate and Comparator Drugs
Description: An adverse event (AE) refers to a treatment-emergent adverse event (TE-AE). A TE-AE is any AE that newly appeared, increased in frequency, or worsened in severity following initiation of study drug.
Time Frame: Up to 40 days (including 30-day follow-up)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 29
Participants | 13 | 3

2. Secondary Outcome: Number of Participants With Investigator's Assessment Indicating Clinical Success at Test of Cure (TOC) Visit (Intent to Treat Analysis Set)
Description: Investigator's assessment of clinical success is defined as (1) resolution or near resolution of most disease-specific signs and symptoms, (2)absence or near resolution of regional or systemic signs of infection (lymphadenopathy, fever, >10% immature neutrophils, abnormal white blood cell count), if present at baseline, and (3) no new signs, symptoms, or complications attributable to the infection under study so no further antibiotic therapy is required for the treatment of the primary lesion.
Time Frame: TOC Visit: 18-25 days after first drug infusion
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 29
Participants | 88 | 27
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Antibiotic Comparator Drug; Test type: Other; Difference in percentages = 3.6, 95% CI 2-sided [-6.3 to 13.5] — The difference (Tedizolid minus Comparator group) in the clinical success rate and 95% confidence interval calculated using the unstratified method of Miettinen and Nurminen

3. Secondary Outcome: Number of Participants With Investigator's Assessment Indicating Clinical Success at TOC Visit (Clinically Evaluable-Test of Cure [CE-TOC] Analysis Set)
Description: as for outcome 2
Time Frame: TOC Visit: 18-25 days after first drug infusion
Population: All randomized participants who received a full dose of study treatment and completed TOC.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 87 | 27
Participants | 87 | 26
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Antibiotic Comparator Drug; Test type: Other; Difference in percentages = 3.7, 95% CI 2-sided [-3.4 to 10.8] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With Early Clinical Responses Measured by Lesion Reduction
Description: Early clinical response is defined as ≥20% reduction from baseline lesion area (defined as length multiplied by the width of the erythema, edema, and/or induration [EEI]) at the 48-72 hour (hr) visit.
Time Frame: 48-72 hr after first drug infusion
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 29
Participants | 84 | 28
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Antibiotic Comparator Drug; Test type: Other; Difference in percentages = -4.2, 95% CI 2-sided [-12.9 to 4.4] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Participants With Investigator's Assessment Indicating Clinical Success at End of Therapy (EOT) Visit (Intent to Treat Analysis Set)
Description: as for outcome 2
Time Frame: EOT Visit: up to 13 days after first drug infusion
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 29
Participants | 88 | 28
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Antibiotic Comparator Drug; Test type: Other; Difference in percentages = 0.2, 95% CI 2-sided [-7.4 to 7.7] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Participants With Investigator's Assessment Indicating Clinical Success at EOT Visit (Clinically Evaluable-End of Therapy [CE-EOT] Analysis Set)
Description: Investigator's assessment of clinical success is defined as (1) resolution or near resolution of most disease-specific signs and symptoms, (2) absence or near resolution of regional or systemic signs of infection (lymphadenopathy, fever, >10% immature neutrophils, abnormal white blood cell count), if present at baseline, and (3) no new signs, symptoms, or complications attributable to the infection under study so no further antibiotic therapy is required for the treatment of the primary lesion.
Time Frame: EOT Visit: up to 13 days after first drug infusion
Population: All randomized participants received a full dose of study treatment and completed EOT.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 87 | 27
Participants | 87 | 27
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Antibiotic Comparator Drug; Test type: Other; Difference in percentages = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 2, analysis 1]

7. Other Pre Specified Outcome: Change From Baseline in Lesion Size
Description: Lesion size is the area in cm^2 of erythema, edema or induration. A negative number corresponds to a decrease in lesion size.
Time Frame: Baseline and TOC visit (18 to 25 days after infusion)
Population: All randomized participants who received a full dose of study treatment, had a baseline value and a TOC visit value (Days 18 to 25).
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 29
cm^2
  Baseline | 135.44 (158.66) | 83.22 (48.55)
  Change at Day 25: number analyzed (Participants) | 88 | 28
  Change at Day 25 | -134.27 (161.18) | -82.51 (49.94)

8. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Tedizolid
Description: The Cmax of tedizolid in plasma after the last dose was estimated based on population pharmacokinetic analysis of observed pharmacokinetic data. Blood samples were collected for pharmacokinetic analysis at specific time points.
Time Frame: Day 1 at 5-80 minutes (min) and 4-12 hrs post-infusion or 2 samples collected between 4-12 hrs after oral dose, at least 60 min apart; at 48-72 hrs: within 60 min prior to administration and 4-12 hrs after administration; and anytime between Day 7 and 9
Population: All randomized participants who received a dose of tedizolid phosphate. Pharmacokinetic analysis was not performed with participants receiving antibiotic comparator drug.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 0
µg/mL | 3.13 [2.89 to 3.38] |

9. Other Pre Specified Outcome: Area Under the Plasma Concentration Versus Time Curve Time 0 to 24 Hours (AUC0-24h) of Tedizolid
Description: AUC0-24h is a measure of the total tedizolid exposure in the plasma from the dose to 24 hours after last dose. AUC0-24h was estimated based on population pharmacokinetic analysis of observed pharmacokinetic data. Blood samples were collected for pharmacokinetic analysis at specific time points.
Time Frame: Day 1 at 5-80 min and 4-12 hrs post-infusion or 2 samples collected between 4-12 hrs after oral dose, at least 60 min apart; at 48-72 hrs: within 60 min prior to administration and 4-12 hrs after administration; and anytime between Day 7 and 9
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: µg*h/mL
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
Number analyzed (Participants) | 91 | 0
µg*h/mL | 28.6 [26.6 to 30.8] |

ADVERSE EVENTS:
Time Frame: Up to 40 days (including 30-day follow-up)
Arm/Group | Tedizolid Phosphate | Antibiotic Comparator Drug
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/91 | 0/29
Other Adverse Events (participants affected / at risk) | 0/91 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid Phosphate (N=91) | Antibiotic Comparator Drug (N=29)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to pursue publication of the results of the study in cooperation with a lead Investigator, subject to the terms and conditions of the clinical study agreement between Sponsor and Investigators. Sponsor approval in writing is required for publication of any data subsets.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT02276482/Prot_SAP_000.pdf